CLINICAL TRIAL: NCT05283551
Title: A Phase 2 Open Label Clinical Trial to Determine the Effect of Famciclovir on Epstein-Barr Virus Activity as Measured by EBV Shedding in Saliva of Patients With Multiple Sclerosis.
Brief Title: Famciclovir in Multiple Sclerosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 249627
Record Dates: First submitted 2022-02-24; First posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-02

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Famciclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: Famciclovir

INTERVENTIONS:
Drug: Famciclovir — Famciclovir (500mg BD)

SUMMARY:
This is a proof-of-concept study in 30 patients with established Relapsing Remitting Multiple Sclerosis (RRMS). IMP is Famciclovir. It is a phase II type A open label study. Each individuals participation in the study will last 36 weeks and will be divided into three phases: pre-treatment (12 weeks), treatment with famciclovir (12 weeks), and post-treatment (12 weeks). During the first 12 week phase patients will remain on their usual treatment alone; this will be followed by three months of co-treatment with famciclovir and then followed by a final three months post-famciclovir treatment where participants will continue to take their usual treatment for RRMS. The primary aim is to explore the effect of famciclovir (500mg BD) on Epstein-Barr virus (EBV) shedding in the saliva of patients with MS

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with MS
* Males and females aged over 18
* Taking Natalizumab (Tysabri) for the treatment of MS,
* Be able to provide informed consent to take part in this study.
* Female patients of childbearing potential (defined in section 13.4) must be willing to follow protocol contraceptive requirements.

Exclusion Criteria:

* Taking MS disease modifying treatment other than natalizumab (Tysabri)
* On no treatment for MS
* Taking additional immunomodulatory agents (either for MS treatment or other reasons)
* Has received a course of high dose oral or intravenous steroids within 3 months of study entry. The use of low dose (total daily dose <10mg) and/or the use of topical steroids will not act as an exclusion criteria.
* Taking antiviral or antiretroviral medication for any reason
* Known allergy to penciclovir, acyclovir, valaciclovir or famciclovir
* Taking probenecid
* Significant renal (CKD 3 or 4) and/or liver (ALT>3x ULN) impairment
* Pregnant, or unwilling to take measures to prevent pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-11-25 (Actual); Primary Completion 2023-11-25 (Estimated); Study Completion 2023-11-25 (Estimated)

PRIMARY OUTCOMES:
Effect of famciclovir on Epstein-Barr virus (EBV) shedding | Baseline to 36 Weeks
  The primary outcome of this study is quantification of Epstein-Barr virus (EBV) shedding in saliva in the IMP treatment phase (famciclovir 500mg BD) and post treatment phase of the Study compared with Epstein-Barr virus (EBV) shedding in saliva in the pre-treatment phase of the Study Shedding is defined as EBV DNA levels in saliva >5.8 copies/ml.

OTHER OUTCOMES:
Explore the effect of famciclovir (500mg BD) on serological markers of Epstein-Barr virus (EBV) infection (anti-EBNA-1 and anti-VCA IgG) | Baseline to 36 Weeks
  Level of serological markers of EBV infection (anti-EBNA-1 IgG and anti-VCA IgG) in particpants' blood in the IMP treatment phase (famciclovir 500mg BD) and post treatment phase of the Study compared with level of serological markers of EBV infection (anti-EBNA-1 IgG and anti-VCA IgG) in the pre-treatment phase of the Study
Explore the effect of famciclovir (500mg BD) on Epstein-Barr virus (EBV) viral replication in blood | Baseline to 36 Weeks
  Level of of EBV DNA in particpants' blood in the IMP treatment phase (famciclovir 500mg BD) and post treatment phase of the Study compared with level of EBV DNA in in the pre-treatment phase of the Study

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dobson R, Holden D, Vickaryous N, Bestwick J, George K, Sayali T, Bianchi L, Wafa M, Gold J, Giovannoni G. A phase 2a open-label clinical trial to determine the effect of famciclovir on EBV activity as measured by EBV shedding in the saliva of patients with multiple sclerosis. Mult Scler. 2024 Jan;30(1):63-70. doi: 10.1177/13524585231215268. Epub 2023 Dec 22. PMID 38131621